CLINICAL TRIAL: NCT06631755
Title: Influence of Vessel Wall Calcification on Early Stent Strut Healing (CaOCT Study)
Brief Title: Influence of Vessel Wall Calcification on Early Stent Strut Healing
Acronym: CaOCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación EPIC (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EPIC41-CaOCT
Record Dates: First submitted 2024-10-02; First posted 2024-10-08 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Coronary Artery Disease
Keywords: Calcification; Strut coverage; Optical Coherence Tomography (OCT)
MeSH Terms: conditions — Coronary Artery Disease; Calcinosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Coronary Artery Disease (CAD) (Other)
  Interventions: Device: Xience Skypoint stent over calcified coronary lesions

INTERVENTIONS:
Device: Xience Skypoint stent over calcified coronary lesions — Patients with Xience Skypoint stent implanted after OCT assesment of calcification

SUMMARY:
To assess the influence of superficial calcium on the early endothelialization (1 month) of the struts of the Xience Skypoint stent (comparing struts with underlying superficial calcium to struts without underlying calcification)

DETAILED DESCRIPTION:
To assess the influence of superficial calcium on the early endothelialization (1 month) of the struts of the Xience Skypoint stent (comparing struts with underlying superficial calcium to struts without underlying calcificatition by opticaL COHERENCE TOMOGRAPHY.

ELIGIBILITY:
Inclusion Criteria:

Patients who meet all the following conditions will be included:

* Patients aged ≥ 18 years old and;
* Patients with clinical indication for stent implantation and;
* Patients with OCT evaluation that shows the presence of calcified tissue underlying the lumen surface, fulfilling the definition of superficial calcium (The distance from the abluminal point of the calcium to the luminal surface is less than 500 μm, in a perpendicular axis to the vessel luminal surface. When referred to the stent struts it will be assumed that such distance of less than 500 μm will be measured between the centre of the abluminal surface of the strut and the abluminal point of the calcium, in the same perpendicular axis).and;
* Patients with good quality baseline OCT evaluation as judged by the investigators and;
* Patients who have been briefed on the study characteristics and have given their prior written informed consent.

Exclusion Criteria:

* Patients who meet, at least, 1 of the following conditions will be excluded:
* Patients with current ST-elevation Myocardial Infarction (STEMI).
* Patients with non-native lesion: stent restenosis, segment previously treated with drug eluting balloon, arterial or saphenous vein grafts.
* Patients with contraindication for the 1-month follow-up angiography and OCT:

  * Glomerular Filtration Rate (GFR)< 30 ml/min/1.72m2
  * Contrast allergy
  * Baseline post-stent control OCT failure, due to tortuosity or any other reason.
* Patient not candidate for a follow up angiography, due to frailty, non-cardiac disease or whatever other condition considered by the local team.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-11-07 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Mean strut coverage thickness of stent | 1 month
  Mean strut coverage thickness (μ) of the stent struts located over superficial calcium will be compared to the mean strut coverage thickness of the struts in the calcium free frames by Optical Coherence Tomography (OCT).

SECONDARY OUTCOMES:
Proportion of covered struts | 1 month
  proportion of covered struts (%) lying over superficial calcium compared to the proportion of covered struts in calcium free frames
Proportion of uncovered struts | 1 month
  Proportion of uncovered struts by OCT at 1 month comparing calcified and non-calcified struts by OCT
Proportion of acute post PCI malapposition struts | 1 month
  Proportion of acute post PCI malapposition comparing calcified and non-calcified struts by OCT
Proportion of malapposed struts | 1 month
  Proportion of malapposed struts comparing calcified and non-calcified struts by OCT at 1 month
Proportion of the resolution of the baseline malapposition struts | 1 month
  Proportion of the resolution of the baseline malapposition struts according to the presence of underlying superficial calcium by OCT at 1 month
Degree of endothelialization | 1 month
  Difference in mean struck coverage thickness between calcified lesion and no calcified lesion
Major adverse cardiovascular events (MACE) | 6 months
  Major adverse cardiovascular events (MACE) defined as a composite of all-cause mortality, cardiac death, myocardial infarction, or target vessel revascularization at 6 months
All Death | 6 months
  Freedom from all Death
Cardiac Death | 6 months
  Freedom from Cardiac Death
Myocardial Infarction | 6 months
  Freedom from Myocardial Infarction
Target Vessel Revascularization | 6 months
  Freedom from Target Vessel Revascularization

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitari Vall Hebron, Barcelona, Spain

REFERENCES:
- [Background] Genereux P, Madhavan MV, Mintz GS, Maehara A, Palmerini T, Lasalle L, Xu K, McAndrew T, Kirtane A, Lansky AJ, Brener SJ, Mehran R, Stone GW. Ischemic outcomes after coronary intervention of calcified vessels in acute coronary syndromes. Pooled analysis from the HORIZONS-AMI (Harmonizing Outcomes With Revascularization and Stents in Acute Myocardial Infarction) and ACUITY (Acute Catheterization and Urgent Intervention Triage Strategy) TRIALS. J Am Coll Cardiol. 2014 May 13;63(18):1845-54. doi: 10.1016/j.jacc.2014.01.034. Epub 2014 Feb 19. PMID 24561145
- [Background] Mosseri M, Satler LF, Pichard AD, Waksman R. Impact of vessel calcification on outcomes after coronary stenting. Cardiovasc Revasc Med. 2005 Oct-Dec;6(4):147-53. doi: 10.1016/j.carrev.2005.08.008. PMID 16326375
- [Background] Lindsay AC, Paulo M, Kadriye K, Tejeiro R, Alegria-Barrero E, Chan PH, Foin N, Syrseloudis D, Di Mario C. Predictors of stent strut malapposition in calcified vessels using frequency-domain optical coherence tomography. J Invasive Cardiol. 2013 Sep;25(9):429-34. PMID 23995714
- [Background] Honda Y, Toyama T, Miyaishi Y, Kan H, Kawaguchi R, Adachi H, Hoshizaki H, Oshima S. Coronary artery calcification as a new predictor of non-target lesion revascularization during the chronic phase after successful percutaneous coronary intervention. Cardiovasc Interv Ther. 2014 Oct;29(4):315-23. doi: 10.1007/s12928-014-0274-4. Epub 2014 Jun 7. PMID 24906449
- [Background] Madhavan MV, Tarigopula M, Mintz GS, Maehara A, Stone GW, Genereux P. Coronary artery calcification: pathogenesis and prognostic implications. J Am Coll Cardiol. 2014 May 6;63(17):1703-14. doi: 10.1016/j.jacc.2014.01.017. Epub 2014 Feb 12. PMID 24530667
- [Background] Otaegui Irurueta I, Gonzalez Sucarrats S, Barron Molina JL, Perez de Prado A, Massotti M, Carmona Ramirez MA, Marti G, Bellera N, Serra B, Serra V, Domingo E, Lopez-Benito M, Sabate M, Ferreira Gonzalez I, Garcia Del Blanco B. Can an ultrathin strut stent design and a polymer free, proendothelializing probucol matrix coating improve early strut healing? The FRIENDLY-OCT trial. An intra-patient randomized study with OCT, evaluating early strut coverage of a novel probucol coated polymer-free and ultra-thin strut sirolimus-eluting stent compared to a biodegradable polymer sirolimus-eluting stent. Int J Cardiol. 2022 Aug 1;360:13-20. doi: 10.1016/j.ijcard.2022.04.043. Epub 2022 Apr 25. PMID 35472561